CLINICAL TRIAL: NCT06954025
Title: High-Intensity Inpatient MDMA-Assisted Psychotherapy for Treatment-Refractory Posttraumatic Stress Disorder: An Open-Label Pilot Study
Brief Title: High-Intensity Inpatient MDMA-Assisted Psychotherapy for PTSD
Acronym: HI-MAP
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: ARQ National Psychotrauma Centre (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HI-MAP
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: MDMA-assisted psychotherapy; Posttraumatic stress disorder; 3,4-Methylenedioxymethamphetamine; Midomafetamine; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDMA-assisted psychotherapy (Experimental): High-intensity MDMA-assisted psychotherapy within an inpatient setting
  Interventions: Drug: High-intensity inpatient MDMA-assisted psychotherapy

INTERVENTIONS:
Drug: High-intensity inpatient MDMA-assisted psychotherapy — Drug: 3,4-methylenedioxymethamphetamine (MDMA) Session 1: 80 mg MDMA HCl followed by a supplemental dose of 40 mg Session 2: 120 mg MDMA HCl followed by a supplemental dose of 60 mg
  Psychotherapy: manualized psychotherapy

SUMMARY:
This study will evaluate the feasibility, safety and efficacy of high-intensity inpatient MDMA-assisted psychotherapy for treatment-refractory posttraumatic stress disorder.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a debilitating condition, which is characterized by re-experiencing, avoidance, and hyperarousal symptoms that have developed following a traumatic experience. Patients suffering from PTSD usually experience a strong negative impact from the disorder on their daily life, diminished cognitive and psychosocial functioning, fractured relationships, inability to maintain employment, substance abuse, high-cost healthcare utilization, increased depression, and suicide risk.

Current evidence-based treatments include trauma-focused therapies (e.g., EMDR and prolonged exposure) and pharmacotherapies (e.g., paroxetine and sertraline). However, PTSD often remains a chronic illness, with high rates of psychiatric and medical comorbidity. One promising new approach involves the use of certain psychoactive drugs as adjuncts to psychotherapy. One drug that has shown particularly promising effects when used within such a substance-assisted therapy approach, is 3,4-methylenedioxymethamphetamine (MDMA). The main rationale behind MDMA-assisted therapy is that MDMA acts as a catalyst to therapy, by reducing the fear response to anxiety provoking stimuli, including previous trauma and traumatic memories. In addition, MDMA enhances introspection and increases interpersonal trust, which can benefit the therapeutic alliance. From a clinical perspective, MDMA alters cognition very slightly, produces only mild sensory alterations, and does not induce a clouding of consciousness, while patients sustain a clear memory of the experience. These subjective effects of MDMA seem to create a productive psychological state that can enhance the therapeutic process.

In the past two decades, several Phase 2 and 3 studies have demonstrated superior efficacy of manualized MDMA-assisted therapy over therapy with placebo or low dose MDMA. These studies provided evidence that chronic PTSD, independent of cause, may be treatable with two to three sessions of MDMA-assisted therapy and associated non-drug preparatory and integrative therapy sessions.

The efficacy and acceptable risk-benefit safety ratio demonstrated in these studies and the potential regulatory approval of this novel therapy, raises several questions, both on how MDMA-assisted therapy could be implemented in national healthcare infrastructures, and on how to tailor the treatment to different PTSD subpopulations. For example, until now MDMA-assisted therapy has solely been studied as an outpatient treatment that takes places over the course of several months. However, a significant percentage of patients with PTSD might benefit from an inpatient setting with an increased frequency of therapy sessions. Several recent studies have investigated such a high intensity inpatient approach to the treatment of PTSD, in which daily trauma focused therapies such as EMDR and prolonged exposure are integrated within a one- to two-week treatment program that includes physical and other activities. In addition to the promising efficacy of this approach, it also offers several other potential benefits, such as increased safety and lower dropout rates. Studying the feasibility of such a high-intensity inpatient approach to MDMA-assisted therapy could broaden its potential future application to a wider range of PTSD subpopulations, including patients with common comorbid conditions that are currently being excluded from MDMA-assisted therapy studies, such as substance use disorders, personality disorders and patients with a higher risk for suicidality. Furthermore, intensifying MDMA-assisted therapy within several weeks of inpatient treatment, might also further increase its efficacy and higher the probability of long-term durability of its effects on PTSD symptoms, by optimizing the integration process in the days and weeks following MDMA sessions.

This open-label pilot study aims to gather supportive data on the feasibility, safety and efficacy of such a High-Intensity approach to delivering MDMA-assisted therapy (HI-MAP). As an initial pilot study, it will focus on a population of treatment-refractory PTSD patients with current moderate to severe PTSD which did not benefit from at least two evidence-based psychotherapies (e.g., EMDR and Prolonged Exposure) for PTSD. This corresponds with the current Dutch standard of care, which recommends to intensify treatment at this stage. Two Experimental Sessions of manualized MDMA-assisted therapy spaced two weeks apart will be integrated within a four-week inpatient treatment program, with preparatory and integrative therapy. The study will be conducted at ARQ Centre'45, a specialized PTSD treatment center, which has been offering high intensity inpatient treatments for years and which has also functioned as a primary study site in a multisite European Phase 2 study into the effects of outpatient MDMA-assisted therapy for the treatment of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Able to provide written informed consent.
* Fluent in speaking and reading Dutch.
* Able to swallow pills.
* Body weight of at least 48 kg.
* Meet DSM-5 criteria for current PTSD.
* Meet criteria for treatment-refractory PTSD.
* Currently in treatment at ARQ Centre'45.
* Agree to have study visits audiovisually recorded.
* Able to provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of the participant becoming unwell or unreachable.

Exclusion Criteria:

* Has a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate.
* Has uncontrolled hypertension.
* Has a recent history of clinically significant hyponatremia or hyperthermia.
* Has current unstable liver or biliary disease.
* Unable or unwilling to safely taper-off prohibited psychiatric medication.
* Has engaged in a new form of psychiatric or mental health care within 12 weeks of enrollment, including Electroconvulsive Therapy (ECT).
* Has a medical or psychiatric condition that could interfere with study participation or pose a risk to the participant's safety or well-being.
* Has any current problem which, in the opinion of the investigator, might interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R) | From Baseline to 1 month after final integrative psychotherapy session
  The last month CAPS-5-R is a semi-structured interview that assesses index history of DSM-5-defined traumatic event exposure, including the most distressing event and time since exposure, to produce a diagnostic score (presence vs. absence) and a PTSD Total Severity score. The CAPS-5-R rates intrusion symptoms (intrusive thoughts or memories), avoidance, cognitive and mood symptoms, arousal and reactivity symptoms, duration and degree of distress and dissociation. The CAPS-5-R will be administered by a study independent CAPS rater.

SECONDARY OUTCOMES:
Sheehan Disability Scale | From Baseline to 1 month after final integrative psychotherapy session
  The Sheehan Disability Scale is a 3-item assessment of functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- ARQ National Psychotrauma Centre / ARQ Centrum'45, Oegstgeest, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Woudenberg C, Voorendonk EM, Bongaerts H, Zoet HA, Verhagen M, Lee CW, van Minnen A, De Jongh A. Effectiveness of an intensive treatment programme combining prolonged exposure and eye movement desensitization and reprocessing for severe post-traumatic stress disorder. Eur J Psychotraumatol. 2018 Jul 10;9(1):1487225. doi: 10.1080/20008198.2018.1487225. eCollection 2018. PMID 30013726
- [Background] Zepeda Mendez M, Nijdam MJ, Ter Heide FJJ, van der Aa N, Olff M. A five-day inpatient EMDR treatment programme for PTSD: pilot study. Eur J Psychotraumatol. 2018 Feb 5;9(1):1425575. doi: 10.1080/20008198.2018.1425575. eCollection 2018. PMID 29441152
- [Background] Feduccia AA, Jerome L, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Breakthrough for Trauma Treatment: Safety and Efficacy of MDMA-Assisted Psychotherapy Compared to Paroxetine and Sertraline. Front Psychiatry. 2019 Sep 12;10:650. doi: 10.3389/fpsyt.2019.00650. eCollection 2019. PMID 31572236
- [Background] Mitchell JM, Ot'alora G M, van der Kolk B, Shannon S, Bogenschutz M, Gelfand Y, Paleos C, Nicholas CR, Quevedo S, Balliett B, Hamilton S, Mithoefer M, Kleiman S, Parker-Guilbert K, Tzarfaty K, Harrison C, de Boer A, Doblin R, Yazar-Klosinski B; MAPP2 Study Collaborator Group. MDMA-assisted therapy for moderate to severe PTSD: a randomized, placebo-controlled phase 3 trial. Nat Med. 2023 Oct;29(10):2473-2480. doi: 10.1038/s41591-023-02565-4. Epub 2023 Sep 14. PMID 37709999
- [Background] Mitchell JM, Bogenschutz M, Lilienstein A, Harrison C, Kleiman S, Parker-Guilbert K, Ot'alora G M, Garas W, Paleos C, Gorman I, Nicholas C, Mithoefer M, Carlin S, Poulter B, Mithoefer A, Quevedo S, Wells G, Klaire SS, van der Kolk B, Tzarfaty K, Amiaz R, Worthy R, Shannon S, Woolley JD, Marta C, Gelfand Y, Hapke E, Amar S, Wallach Y, Brown R, Hamilton S, Wang JB, Coker A, Matthews R, de Boer A, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted therapy for severe PTSD: a randomized, double-blind, placebo-controlled phase 3 study. Nat Med. 2021 Jun;27(6):1025-1033. doi: 10.1038/s41591-021-01336-3. Epub 2021 May 10. PMID 33972795